CLINICAL TRIAL: NCT05541484
Title: Ketone Monitoring in T1D: Effect of SGLT2i During Usual Care and With Insulin Deficiency
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: Juvenile Diabetes Research Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 202206078
Record Dates: First submitted 2022-09-12; First posted 2022-09-15 (Actual); Results first posted 2025-02-21 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2025-01

CONDITIONS: Diabetes Mellitus, Type 1
Keywords: ketosis; beta hydroxybutyrate; sodium glucose co-transport inhibitor; breath ketone
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Ketosis | interventions — Sodium-Glucose Transporter 2 Inhibitors; dapagliflozin

STUDY DESIGN:
Intervention Model Description: Participants will test the breath ketone analyzer under usual care or with usual care plus SGLT2i treatment. Each out patient segment will last two weeks. At the end of each out patient segment, participants will undergo a one-day insulin withdrawal period with more intense monitoring.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Usual care (UC) or Dapagliflozin (DAPA) (Other): 20 persons with T1D
  Interventions: Drug: SGLT2 inhibitor; Device: Biosense Breath Ketone Analyzer

INTERVENTIONS:
Drug: SGLT2 inhibitor — See above.
  Other Names: Dapagliflozin 10mg (Farxiga)
Device: Biosense Breath Ketone Analyzer — The hand-held device tests ketones in exhaled breath

SUMMARY:
This proposed study will test whether measurement of breath acetone (BrAce) can be used for the purpose of identifying ketosis (elevated ketones) in persons with type 1 diabetes (T1D). This is important for the potential use of sodium glucose co-transport inhibitors (SGLT2i) in persons with T1D.

DETAILED DESCRIPTION:
The study will consist of 4 distinct segments that include routine testing of ketones during usual care, during insulin deficiency, and while taking a SGLT2i in addition to usual care, then with insulin deficiency after the SGLT2i has reached steady state and ingested that morning, in a crossover design. We will study 20 adults with T1D who are using Dexcom G6 continuous glucose monitor (CGM), plus any form of insulin delivery. Simultaneous ketone monitoring using a the Biosense® breath ketone analyzer (BKA) and capillary blood beta hydroxybutyrate (BOHB) measurement will be done 2-3 times daily for 2 weeks during each of the outpatient segments. This will generate > 800 data points comparing breath acetone, measured in units called ACEs, versus capillary blood BOHB measurements for each 2 week period. On days of insulin withdrawal, which will take place on the Washington University Intensive Research Unit (IRU), frequent monitoring with capillary blood measurements of BOHB (Precision Xtra®, Abbott) will be compared with breath BrAce measurements (Biosense®, Readout) and laboratory measurements of BOHB and acetoacetate. Electrolytes and glucose will also be measured.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 diabetes for >1 year
* Age 18 - 75, any gender, race or ethnicity
* HbA1c <10%
* Stable insulin delivery method for the past 30 days
* Vision of 20/40 or better, including ability to read all device instructions and insulin pump settings
* Use of an insulin pump and ability to make adjustments to pump settings
* Insulin delivery by MDI with basal insulin (glargine U100) given in the morning OR willingness to transition to basal glargine given in the morning for at least 48 hours prior to insulin withdrawal visits
* Use of personal CGM, only Dexcom G6 will be permitted for data consistency
* Use of cellular phone (iOS11 and above or Android) with data capability with connectivity to Dexcom Clarity app and Biosense Ketone Monitoring app
* Willing to share CGM, capillary ketone results and BrACE data with the study group
* Able to understand the study requirements, risks and benefits and able to provide written informed consent
* Able to schedule the visits and perform study related tasks

Exclusion Criteria:

* History of DKA in the past 6 months, or more than 1 episode of DKA in the past 2 years
* Use of insulin degludec, insulin glargine U300 or insulin detemir as basal insulin and unwilling to transition to glargine given in the morning for at least 48 hours before the insulin withdrawal visits
* Use of an SGLT2i in the past 30 days or intolerance to SGLT2i use in the past for any reason
* Unstable heart disease, including hospitalization for any cardiac or vascular event in the past 6 months.
* eGFR <30 ml/min/1.73m2 or hemoglobin <11.0 g/dL measured in the past year
* Cancer that has been under treatment in the past 6 months, or treatment is likely in the 3 months after signing the consent, not including skin cancer or cancers under long-term hormonal reduction treatment (breast or prostate, no other active treatment)
* Psychiatric condition that interferes with daily activities or diabetes self-care, including substance abuse
* Any illness or condition that may interfere with study measurements, or contraindications for use of SGLT2i, based on investigator discretion (hemoglobinopathy, orthostatic hypotension)
* Unwilling to avoid alcohol during the active study periods, specifically to avoid alcohol for 4 hours prior to any breath ketone measurement
* Currently following or planning to adopt a diet that is low in carbohydrates (defined as <90 grams of carbohydrate per day) or is expected to be ketogenic
* Use of oral or injected corticosteroids within the past 30 days or planned during the study period
* Taking disulfiram (due to interference with breath ketone measurements)
* History of vomiting episodes for any reason in the past 30 days, or hospitalization for cyclic vomiting in the past year
* History of urinary tract infection in the past 3 months
* Pregnancy, breast-feeding or intention of becoming pregnant during the study time period and up to 30 days after study completion
* Pre-menopausal women not using acceptable birth control defined as abstinence, surgical sterilization, hysterectomy, hormonal contraception, IUD or proven effective barrier methods

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2022-10-14 (Actual); Primary Completion 2023-12-23 (Actual); Study Completion 2023-12-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janet B McGill, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: Undecided
After all analyses have been completed and papers have been published, the investigators plan to share the IPD. Detailed plan will be forthcoming.

REFERENCES:
- [Background] Dandona P, Mathieu C, Phillip M, Hansen L, Griffen SC, Tschope D, Thoren F, Xu J, Langkilde AM; DEPICT-1 Investigators. Efficacy and safety of dapagliflozin in patients with inadequately controlled type 1 diabetes (DEPICT-1): 24 week results from a multicentre, double-blind, phase 3, randomised controlled trial. Lancet Diabetes Endocrinol. 2017 Nov;5(11):864-876. doi: 10.1016/S2213-8587(17)30308-X. Epub 2017 Sep 14. PMID 28919061
- [Background] Mathieu C, Dandona P, Gillard P, Senior P, Hasslacher C, Araki E, Lind M, Bain SC, Jabbour S, Arya N, Hansen L, Thoren F, Langkilde AM; DEPICT-2 Investigators. Efficacy and Safety of Dapagliflozin in Patients With Inadequately Controlled Type 1 Diabetes (the DEPICT-2 Study): 24-Week Results From a Randomized Controlled Trial. Diabetes Care. 2018 Sep;41(9):1938-1946. doi: 10.2337/dc18-0623. Epub 2018 Jul 19. PMID 30026335
- [Background] Owen OE, Trapp VE, Skutches CL, Mozzoli MA, Hoeldtke RD, Boden G, Reichard GA Jr. Acetone metabolism during diabetic ketoacidosis. Diabetes. 1982 Mar;31(3):242-8. doi: 10.2337/diab.31.3.242. PMID 6818074
- [Background] Garg SK, Peters AL, Buse JB, Danne T. Strategy for Mitigating DKA Risk in Patients with Type 1 Diabetes on Adjunctive Treatment with SGLT Inhibitors: A STICH Protocol. Diabetes Technol Ther. 2018 Sep;20(9):571-575. doi: 10.1089/dia.2018.0246. Epub 2018 Aug 21. No abstract available. PMID 30129772
- [Background] Laffel L. Ketone bodies: a review of physiology, pathophysiology and application of monitoring to diabetes. Diabetes Metab Res Rev. 1999 Nov-Dec;15(6):412-26. doi: 10.1002/(sici)1520-7560(199911/12)15:63.0.co;2-8. PMID 10634967
- [Background] Hancock G, Sharma S, Galpin M, Lunn D, Megson C, Peverall R, Richmond G, Ritchie GAD, Owen KR. The correlation between breath acetone and blood betahydroxybutyrate in individuals with type 1 diabetes. J Breath Res. 2020 Oct 29;15(1):017101. doi: 10.1088/1752-7163/abbf37. PMID 33027776
- [Background] Suntrup Iii DJ, Ratto TV, Ratto M, McCarter JP. Characterization of a high-resolution breath acetone meter for ketosis monitoring. PeerJ. 2020 Sep 24;8:e9969. doi: 10.7717/peerj.9969. eCollection 2020. PMID 33024634
- [Background] Spanel P, Dryahina K, Rejskova A, Chippendale TW, Smith D. Breath acetone concentration; biological variability and the influence of diet. Physiol Meas. 2011 Aug;32(8):N23-31. doi: 10.1088/0967-3334/32/8/N01. Epub 2011 Jul 1. PMID 21725144
- [Background] Rydosz A. A Negative Correlation Between Blood Glucose and Acetone Measured in Healthy and Type 1 Diabetes Mellitus Patient Breath. J Diabetes Sci Technol. 2015 Jul;9(4):881-4. doi: 10.1177/1932296815572366. Epub 2015 Feb 17. PMID 25691653
- [Background] Herring RA, Shojaee-Moradie F, Garesse R, Stevenage M, Jackson N, Fielding BA, Mendis A, Johnsen S, Umpleby AM, Davies M, Russell-Jones DL. Metabolic Effects of an SGLT2 Inhibitor (Dapagliflozin) During a Period of Acute Insulin Withdrawal and Development of Ketoacidosis in People With Type 1 Diabetes. Diabetes Care. 2020 Sep;43(9):2128-2136. doi: 10.2337/dc19-2579. Epub 2020 Jul 8. PMID 32641376
- [Background] Patel NS, Van Name MA, Cengiz E, Carria LR, Weinzimer SA, Tamborlane WV, Sherr JL. Altered Patterns of Early Metabolic Decompensation in Type 1 Diabetes During Treatment with a SGLT2 Inhibitor: An Insulin Pump Suspension Study. Diabetes Technol Ther. 2017 Nov;19(11):618-622. doi: 10.1089/dia.2017.0267. Epub 2017 Oct 25. PMID 29068709
- [Derived] Jones KE, Petersen MC, Markov AM, Salam M, Krutilova P, McKee AM, Bohnert KL, Adamson SE, McGill JB. Breath Acetone Correlates With Capillary beta-hydroxybutyrate in Type 1 Diabetes. J Diabetes Sci Technol. 2025 Apr 22:19322968251334640. doi: 10.1177/19322968251334640. Online ahead of print. PMID 40260699
- [Derived] Jones KE, Petersen MC, Markov AM, Salam M, Krutilova P, McKee AM, Bohnert KL, Adamson SE, McGill JB. Breath Acetone Correlates with Capillary beta-hydroxybutyrate in Type 1 Diabetes. medRxiv [Preprint]. 2025 Jan 31:2025.01.30.25321320. doi: 10.1101/2025.01.30.25321320. PMID 39974120

RESULTS

PARTICIPANT FLOW:
Groups:
- Group A: Usual Care Followed by Usual Care Plus Dapagliflozin: 10 persons with T1D will check capillary beta hydroxybutyrate (BOHB) and concomitant breath acetone (BrAce) 2 - 3 times daily for 2 weeks during usual care, then undergo an insulin withdrawal visit. Subsequently, the Group A patients will repeat the paired measurements of BOHB and BrAce, 2 - 3 times daily for 2 weeks during usual care plus treatment with the SGLT2i dapagliflozin, 10 mg taken orally daily, followed by an insulin withdrawal visit.
  SGLT2 inhibitor: See above.
  Biosense Breath Ketone Analyzer: The hand-held device tests ketones in exhaled breath
- Group B: Usual Care Plus Dapagliflozin Followed by Usual Care: 10 persons with T1D will check capillary beta hydroxybutyrate (BOHB) and concomitant breath acetone (BrAce) 2 - 3 times daily for 2 weeks during usual care plus treatment with the SGLT2i dapagliflozin, 10 mg taken orally daily, then undergo an insulin withdrawal visit. Subsequently, the Group B patients will repeat the paired measurements of BOHB and BrAce, 2 - 3 times daily during usual care alone followed by an insulin withdrawal visit.
  SGLT2 inhibitor: See above.
  Biosense Breath Ketone Analyzer: The hand-held device tests ketones in exhaled breath
Period: Overall Study
Arm/Group | Group A: Usual Care Followed by Usual Care Plus Dapagliflozin | Group B: Usual Care Plus Dapagliflozin Followed by Usual Care
Started | 11 | 10
Completed | 10 | 10
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Population: same
Arm/Group | Usual Care (UC) or Dapagliflozin (DAPA)
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 13
  >=65 years | 7
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.0 (18.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 11
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 19
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: Capillary Blood Beta-hydroxybutyrate (BOHB) During Outpatient Care
Description: Differences between usual care v dapagliflozin of capillary beta hydroxybutyrate (BOHB) measurements during outpatient care.
Time Frame: Measurements were taken 2-3 times daily for 2 weeks
Measure: Mean (Inter-Quartile Range); unit: mmol/L
Units Other Than Participants: measurements
Groups:
- Usual Care: Two weeks of outpatient care measurements
- Dapagliflozin: Two weeks of outpatient care measurements while taking dapagliflozin
Arm/Group | Usual Care | Dapagliflozin
Number analyzed (Participants) | 20 | 20
Number analyzed (measurements) | 718 | 707
mmol/L | 0.1 [0.1 to 0.2] | 0.2 [0.1 to 0.3]
Statistical Analysis 1: Comparison: Usual Care vs Dapagliflozin; Test type: Other — Spearman's ρ given non-normal variable distributions; p < 0.0001, Wilcoxon (Mann-Whitney) — Spearman's ρ given non-normal variable distributions

2. Primary Outcome: Breath Acetone (BrACE) During Outpatient Care
Description: Differences of breath acetone (BrACE) measurements between usual care v dapagliflozin during outpatient care.
Time Frame: Measurements were taken 2-3 times daily for 2 weeks
Measure: Mean (Inter-Quartile Range); unit: AU (ppm)
Arm/Group | Usual Care | Dapagliflozin
Number analyzed (Participants) | 20 | 20
AU (ppm) | 1 [1 to 3] | 2 [1 to 4]

3. Other Pre Specified Outcome: Ketone Levels in Persons With T1D Undergoing Insulin Withdrawal
Description: Comparison of ketone levels (BOHB and BrAce) during insulin withdrawal after usual care and during insulin withdrawal after usual care plus treatment with an SGLT2i.
Time Frame: 2 days
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: two weeks of outpatient care
Description: Adverse event and/or serious adverse event uses the same definition as clinicaltrials.gov
Groups:
- Usual Care: 20 persons with T1D will check capillary beta hydroxybutyrate (BOHB) and concomitant breath acetone (BrAce) 2 - 3 times daily for 2 weeks during usual care, then undergo an insulin withdrawal visit.
  Biosense Breath Ketone Analyzer: The hand-held device tests ketones in exhaled breath
- Usual Care Plus Dapagliflozin (Dapagliflozin): 20 persons with T1D will check capillary beta hydroxybutyrate (BOHB) and concomitant breath acetone (BrAce) 2 - 3 times daily for 2 weeks during usual care plus treatment with the SGLT2i dapagliflozin, 10 mg taken orally daily, then undergo an insulin withdrawal visit.
  Biosense Breath Ketone Analyzer: The hand-held device tests ketones in exhaled breath
Arm/Group | Usual Care | Usual Care Plus Dapagliflozin (Dapagliflozin)
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 1/20 | 8/20
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Usual Care (N=20) | Usual Care Plus Dapagliflozin (Dapagliflozin) (N=20)
nausea (Endocrine disorders) | 0 (0) | 4 (4)
hypoglycemia (Endocrine disorders) | 0 (0) | 4 (4)
palpitations (Cardiac disorders) | 0 (0) | 1 (1)
gastroenteritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
hyperglycemia (Endocrine disorders) | 1 (1) | 0 (0)
fatigue (Endocrine disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-01-10): https://cdn.clinicaltrials.gov/large-docs/84/NCT05541484/Prot_SAP_000.pdf